CLINICAL TRIAL: NCT01184053
Title: A Phase II Trial of Trisenox in Women With Recurrent or Metastatic Endometrial Adenocarcinoma
Brief Title: Trisenox® in Women With Metastatic Endometrial Cancer
Acronym: NRR
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Accrual was very low. No subject had been enrolled in a year.
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: Cephalon (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCCC 0920
Record Dates: First submitted 2010-07-22; First posted 2010-08-18 (Estimated); Results first posted 2017-06-14 (Actual); Last update posted 2017-06-14 (Actual); Status verified 2017-05

CONDITIONS: Endometrial Carcinoma
Keywords: endometrial; carcinoma; recurrent; metastatic; Trisenox; arsenic trioxide; Phase II; VEGF; gynecology; Lineberger; UNC; vascular endothelial growth factor; University of North Carolina at Chapel Hill
MeSH Terms: conditions — Endometrial Neoplasms; Carcinoma; Recurrence; Neoplasm Metastasis | interventions — Arsenic Trioxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Trisenox treatment (Experimental): Arsenic trioxide - 0.25 mg/kg/day for 5 consecutive days, every 4 weeks.
  Interventions: Drug: Arsenic trioxide

INTERVENTIONS:
Drug: Arsenic trioxide — Arsenic trioxide - 0.25 mg/kg/day for 5 consecutive days, every 4 weeks.
  Other Names: Trisenox

SUMMARY:
The primary purpose of this study is to see whether women who have already received chemotherapy for their endometrial cancer, or who have disease that has spread outside of the uterus, will respond to the drug arsenic trioxide (Trisenox®) as judged by shrinkage of their tumor.

DETAILED DESCRIPTION:
This is an open-label, single arm, single institution, phase II trial designed to assess the response rate and safety of Trisenox® in women with recurrent endometrial carcinoma. Trisenox® will be administered at a dose of 0.25 mg/kg/day for 5 consecutive days (D1-5) every 4 weeks. A 4-week period will be defined as a cycle of treatment. Marker and non-marker lesions will be assessed every 2 cycles (every 8 weeks) and the response assigned according to Gynecologic Oncology Group (GOG) RECIST guidelines. Safety will be assessed by routine physical, laboratory and ECG evaluations. Up to 10 patients will be enrolled into the study. Patients are expected (excluding any unforeseen toxicities) to receive a minimum of 2 and a maximum of 6 cycles of Trisenox®. (Patients with at least documented stable disease may be eligible for >6 cycles). Patients will be followed for 6 months after their last dose of Trisenox®.

For this trial we would allow one prior cytotoxic regimen since the time of recurrence and patients may have had one prior regimen as part of their induction chemotherapy. Patients will be treated with 0.25 mg/kg/day for days 1-5 every 28 days and patients may remain on trial until progression of disease.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years of age with histologically confirmed metastatic or recurrent endometrial cancer
2. Documented progression of their endometrial cancer (i.e., within the last 3 months)
3. If of childbearing potential they must agree to use approved barrier methods of contraception
4. Presence of at least one measurable lesion that:

   * Can be accurately measured in at least one dimension with longest diameter ≥20 mm using conventional techniques or ≥10 mm with spiral CT scan (or otherwise at least twice the reconstruction interval for CT or MRI scans).
   * Previously irradiated lesions may be considered to be measurable provided: 1) there has been documented progression of the lesion(s) since completion of radiotherapy, and 2) the criteria for measurability as outlined above are met.
5. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
6. Minimum life expectancy of 3 months
7. Adequate renal and hepatic function (per study protocol guidelines)
8. Adequate bone marrow function (per study protocol guidelines)
9. Serum cholesterol <350 mg/dL and triglycerides < 400 mg/dL
10. Able to understand and give written informed consent
11. Ejection fraction >55% with no focal left ventricular wall motion abnormalities in patients with a history of coronary artery disease or a history of congestive heart failure.

Exclusion Criteria:

1. Women who are pregnant or lactating
2. Presence of brain metastases
3. Two or more prior cycles of cytotoxic chemotherapy since recurrence (Two total regimens are allowed if one includes adjuvant therapy.)
4. Prior therapy with Trisenox or known sensitivity to this agent
5. Prior anticancer treatment (chemotherapy, radiotherapy, immunotherapy, biological response modifiers, signal transduction inhibitors, etc) within 4 weeks prior to the first dose of Trisenox.
6. Ongoing toxicity associated with prior anticancer therapy (except peripheral neuropathy of ≤ grade 1 by NCI toxicity criteria)
7. Another primary malignancy within the past three years (except for non-melanoma skin cancer and cervical carcinoma in situ)
8. Significant uncontrolled cardiovascular disease
9. Active infection requiring systemic therapy
10. Known HIV infection
11. Treatment with any investigational agent within 4 weeks prior to the first dose of Trisenox
12. Concurrent treatment with immunosuppressive agents other than prescribed corticosteroids
13. Inadequate recovery from any prior surgical procedure or having undergone any major surgical procedure within 2 weeks prior to the first dose of Trisenox
14. Patients having undergone recent placement of a central venous access port will be considered eligible if they have recovered
15. Presence of any other life-threatening illness or organ system dysfunction which, in the opinion of the Investigator, would either compromise the patient's safety or interfere with evaluating the safety of the study drug
16. Prolonged absolute corrected QT interval (QTc) interval > 500 msec
17. Underlying conduction disease that prevents measurement of QT interval
18. History of ventricular tachycardia or any cardiac arrhythmia requiring the placement of an automated intraventricular cardiac defibrillator.
19. Inability to discontinue therapy with class I or class III antiarrhythmic medications.
20. Inability to discontinue drugs known to be associated with a risk for torsades de pointes

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2010-03; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paola Gehrig, MD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (1):
- North Carolina Cancer Hosptial, UNC, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: web address for Lineberger Comprehensive Cancer Center, UNC — http://www.unclineberger.org
- See also: web address for the National Cancer Institute (NCI) — http://www.cancer.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Women 18 years of age with histologically confirmed metastatic or recurrent endometrial cancer at the Lineberger Comprehensive Cancer Center
Period: Overall Study
Arm/Group | Trisenox Treatment
Started | 3
Completed | 0
Not Completed | 3
Not completed — progression while on treatment | 3

BASELINE CHARACTERISTICS:
Arm/Group | Trisenox Treatment
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Objective Response (CR+PR) Rate of Subjects Given Trisenox
Description: To estimate the objective response (CR+PR) rate (as defined by the Gynecologic Oncology Group [GOG] RECIST Criteria)of Trisenox® in women with recurrent or metastatic endometrial cancer when administered at 0.25 mg/kg/day for 5 consecutive days (D1-5) every 4 weeks.
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Trisenox Treatment
Number analyzed (Participants) | 3
Participants | 0

2. Secondary Outcome: Progression Free Survival in Patients Treated With Trisenox®
Description: Progression-Free survival is the period from start of treatment until disease progression, death, or date of last contact.
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Trisenox Treatment
Number analyzed (Participants) | 3
Participants | 0

3. Secondary Outcome: Overall Survival
Time Frame: 5 years
Population: All patients who received treatment
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Trisenox Treatment
Number analyzed (Participants) | 3
days | 320 [59 to NA] — The upper limit of the 95% Confidence Interval was calculated as infinity (and thus NA) due to few events at the time of analysis.

4. Secondary Outcome: Associations Between Markers of Angiogenesis (e.g. VEGF) With Response
Description: We will request a blood sample to measure vascular endothelial growth factor (VEGF) as well as other angiogenic factors and correlate levels to response to arsenic trioxide. Such effects have been observed in cultured cell lines and animal models, as well as clinical studies.
Time Frame: 4 years
Population: No patients achieved a CR or PR response, no angiogenesis was performed.
Arm/Group | Trisenox Treatment
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Trisenox Treatment
All-Cause Mortality (participants affected / at risk) | 2/3
Serious Adverse Events (participants affected / at risk) | 2/3
Other Adverse Events (participants affected / at risk) | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Trisenox Treatment (N=3)
Rapid weight gain (Metabolism and nutrition disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Trisenox Treatment (N=3)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 1 (1)
Ascites (non-malignant) (Gastrointestinal disorders) | 1 (1)
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Creatinine (Investigations) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Edema: limb (General disorders) | 1 (2)
Edema: trunk/genital (General disorders) | 1 (2)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 1 (2)
Flushing (Vascular disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 2 (2)
Insomnia (Psychiatric disorders) | 2 (2)
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 1 (1)
Nail changes (Skin and subcutaneous tissue disorders) | 1 (1)
Pain - Back (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain - Extremity-limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain - Head/headache (Nervous system disorders) | 1 (1)
Pain - Throat/pharynx/larynx (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Palpitations (Cardiac disorders) | 1 (1)
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 1 (1)
Pruritus/itching (Skin and subcutaneous tissue disorders) | 1 (1)
Pulmonary/Upper Respiratory - Other (Specify, __) (Respiratory, thoracic and mediastinal disorders) | 1 (1) — difficulty taking deep breaths
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 1 (1)
Supraventricular and nodal arrhythmia - Sinus tachycardia (Cardiac disorders) | 1 (2)
Thrombosis/thrombus/embolism (Vascular disorders) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Urinary frequency/urgency (Renal and urinary disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
The study accrued few patients secondary to the strict entry criteria regarding labs, EKG, etc in a sick endometrial cancer population.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes